CLINICAL TRIAL: NCT06434519
Title: Evaluation of the Effect of Moisturizers on the Absorption of Metronidazole Into the Stratum Corneum of Rosacea Patients With Tape Stripping and Liquid Chromatography-mass Spectrometry
Brief Title: Metronidazole SC Penetrance With Moisturizers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Rosacea Society (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00114776
Record Dates: First submitted 2024-05-16; First posted 2024-05-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-09

CONDITIONS: Rosacea, Erythematotelangiectatic
Keywords: rosacea; metronidazole; LC-MS; tape strip
MeSH Terms: conditions — Rosacea

STUDY DESIGN:
Intervention Model Description: 5 patients will enrolled in 4 study arms. Each study arm will represent a different combination of moisturizer applied to the face, followed by metronidazole cream. No moisturizer will be applied to the left side of each patient's face, permitting for each patient to represent their own negative (no metronidzole cream applied) and positive control (metronidazole cream + no moisturizer). Metronidazole penetrance in the stratum corneum will be assess with tape strips and LC-MS
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Metronidazole cream + Cetaphil moisturizer (Experimental): Apply Cetaphil (glycerin (humectant) and petrolatum (occlusive)) moisturizer followed by metronidazole cream. Tape striping will occur at 1 hours and 4 hours post metronidazole application.
  Interventions: Drug: Metronidazole cream; Other: Cetaphil moisturizer
- Metronidzole cream + CeraVe moisturizer (Experimental): Apply CeraVe (glycerin/hyaluronic acid (humectant), ceramides (intercellular lipid component), and dimethicone/petrolatum (occlusive)) moisturizer followed by metronidazole cream. Tape striping will occur at 1 hours and 4 hours post metronidazole application.
  Interventions: Drug: Metronidazole cream; Other: CeraVe moisturizer
- Metronidzole cream + Eucerin Healing Lotion moisturizer (Experimental): Apply Eucerin Healing Lotion (mineral oil (occlusive) and sorbitol/propylene glycol (humecants)) followed by metronidazole cream. Tape striping will occur at 1 hours and 4 hours post metronidazole application.
  Interventions: Drug: Metronidazole cream; Other: Eucerin Healing Lotion moisturizer
- Metronidazole cream + Aveeno Calm and Restore Oat Gel moisturizer (Experimental): Apply Aveeno Calm and Restore Oat Gel (glycerin (humectant) and dimethicone (occlusive) and oat kernel flour based gel moisturizer) moisturizer followed by metronidazole cream. Tape striping will occur at 1 hours and 4 hours post metronidazole application.
  Interventions: Drug: Metronidazole cream; Other: Aveeno Calm and Restore Oat Gel moisturizer

INTERVENTIONS:
Drug: Metronidazole cream — After application of one of the moisturizers under investigation in this study to the right side of the patient's face, x5 tape strips will be collected from the left side of a patient's face. These will provide negative controls for quantitation of metronidazole in the stratum corneum. Then, 0.5 mL of a 1% metronidazole cream will be applied to both the right and left sides of a patient's face with clean gloves to prevent cross contamination. Tapes strips x5 will subsequently be collected from the left and right sides of the face at 1 hour and 4 hour time points to assess penetrance of metronidazole through the stratum corneum.
Other: Cetaphil moisturizer — 0.5 mL of moisturizer will be dispensed using a pre-loaded syringe applied to the right face of each patient the patient's standard practice. No moisturizer will be applied to the left side of the face to provide for negative and positive tape strip controls to assess metronidazole penetrance through the stratum corneum in the presence of the moisturizer.
  Arms: Metronidazole cream + Cetaphil moisturizer
Other: CeraVe moisturizer — 0.5 mL of moisturizer will be dispensed using a pre-loaded syringe applied to the right face of each patient the patient's standard practice. No moisturizer will be applied to the left side of the face to provide for negative and positive tape strip controls to assess metronidazole penetrance through the stratum corneum in the presence of the moisturizer.
  Arms: Metronidzole cream + CeraVe moisturizer
Other: Eucerin Healing Lotion moisturizer — 0.5 mL of moisturizer will be dispensed using a pre-loaded syringe applied to the right face of each patient the patient's standard practice. No moisturizer will be applied to the left side of the face to provide for negative and positive tape strip controls to assess metronidazole penetrance through the stratum corneum in the presence of the moisturizer.
  Arms: Metronidzole cream + Eucerin Healing Lotion moisturizer
Other: Aveeno Calm and Restore Oat Gel moisturizer — 0.5 mL of moisturizer will be dispensed using a pre-loaded syringe applied to the right face of each patient the patient's standard practice. No moisturizer will be applied to the left side of the face to provide for negative and positive tape strip controls to assess metronidazole penetrance through the stratum corneum in the presence of the moisturizer.
  Arms: Metronidazole cream + Aveeno Calm and Restore Oat Gel moisturizer

SUMMARY:
Topical metronidazole is a widely used first line treatment for erythemotelangiectatic and inflammatory rosacea. Commonly, a moisturizer is also used to restore the skin barrier and reduce inflammation. The purpose of this study is to assess the whether the common practice of applying moisturizer prior to topical metronidazole affects this medication's stratum corneum penetrance in rosacea patients. Participants will have one research office visit that will consist of having a randomly assigned combination of metronidazole and one of four moisturizers applied to their face, followed by non-invasive tape stripping of skin at the 1 hour and 4 hour time points. These tape strip samples will be analyzed with liquid chromatography mass spectrometry (LC-MS) for assessment of metronidazole penetrance in the stratum corneum in the presence of moisturizers. The target population will be rosacea patients in the age range of 18-60 years of age. This study has minimal risks/safety issues as topical metronidazole is an already FDA approved medication with an indication for rosacea and all investigated moisturizers are over-the-counter formulations commonly used within the rosacea patient population. Tape stripping will remove 5 levels of superficial stratum corneum, and will not result in bleeding, scarring, or other prolonged cosmetic disfigurement. Small, transient bruising may result from tape strip collection. The collected samples will have no to minimal biohazard risk, as the collected specimen for analysis will only contain skin scale; samples will be extracted with organic solvents and decontaminated with a 0.2 micron nylon filter prior to analysis on the LC-MS instrumentation.

DETAILED DESCRIPTION:
Rosacea is a debilitating spectrum of disease causing both socially embarrassing erythema and disfiguring rhinophyma. Treatment is challenging and life-long, often requiring clinicians to trial multiple medications, such as azelaic acid, metronidazole, or ivermectin to achieve disease control. The skin of rosacea patients inherently has impaired skin barrier function, resulting in inflammation and hypersensitivity to most therapeutics. Thus, many clinicians encourage patients to augment their topical medications with personal moisturizers to optimize the skin barrier. However, there is limited data to support that moisturizers do not affect drug epidermal penetrance and efficacy. To the investigator's knowledge, only a single trial assessing the effect of moisturizers on skin penetrance of azelaic acid has been published in the English literature. In the era of evidence-based medicine, it is critical to provide either the scientific data to support or to refute this medical dogma. The investigator's proposal addresses this gap in the basic science literature and will provide data to evaluate a long and widely-held dermatologist recommendation for the treatment of rosacea. The investigators anticipate that there may be preferred combinations of medication and moisturizers based upon the matched lipophilicities and other chemical properties of the occlusive agent and therapeutic drug. Identification of such combinations may lead to improved outcomes for those struggling with treatment-resistant rosacea and lead to additional pharmaceutical advances in the treatment of rosacea.

Drug formulation is critical to the successful treatment of dermatologic disease. An active ingredient must diffuse through the stratum corneum (SC) to reach the dermis to achieve its therapeutic effect. In addition to the intrinsic chemical properties of the active compound dictating the kinetics of the diffusion process, chemists tweak a topical formulation's vehicle, emulsifiers, and polymers to enhance drug SC penetrance and overcome the skin's evolutionary role as a barrier to the outside world. The combination of drug with additional topical moisturizers inherently changes the chemical environment that the active drug must diffuse through to reach the dermis. Moisturizers and other topical cosmetics are well established to affect dermal drug and toxin absorption. For example, moisturizers have been demonstrated to enhance dermal penetrance of herbicide 2,4-dichlorophenoxacetic acid in murine models. Similarly, occlusive moisturizers are often applied over steroids to enhance their anti-inflammatory efficacy, presumably through improved epidermal penetration. Increased penetrance is a case-by-case scenario, however, and considerable attention is dedicated to topical formulation to appropriately modulate therapeutic drug penetrance of the SC during the drug design process.

To the investigator's knowledge, the formulation and timing of moisturizer application on drug efficacy in rosacea is understudied. An extensive literature review revealed only a single study addressing this important question for the special case of azelaic acid with an in vitro Franz cell diffusion assay using donated trunk skin biopsies. In this study, a 14C radiolabeled 15% azelaic acid gel was applied to epidermis before or after the application of Dove Lotion, CeraVe Moisturizer Lotion, and Cetaphil Moisturizing Lotion. The penetrance of azelaic acid into the SC was then assessed up to 48 hours post-application using liquid scintillation spectrometry. Azelaic acid SC penetration was not statistically different between the moisturizers or timing of application, although trends towards decreased penetration was noted in 1 of 3 studied moisturizers. There are several limitations to this study. First, azelaic acid occupies a unique chemical space among rosacea therapies. Azelaic acid's lipophilicity (LogP), an important chemical property affecting epidermal drug penetrance, is 1.6 compared with 5.83, 0.0, -0.3 and -0.7 for ivermectin, metronidazole, monocycline, and doxycycline, respectively, suggesting that azelaic acid is between 1.4e2 times more lipophilic to 1.7e4 times less lipophilic than other therapies. Thus, azelaic acid is a poor standard with which to assess moisturizers' impact on SC drug penetrance. Second, truncal skin was used to assess azelaic acid SC penetrance. Consequently, the study's clinical relevance is limited as rosacea exclusively affects the face, where the skin is much thinner and transdermal absorption occurs more readily. Finally, although a tritium diffusion control was implemented to select skin samples with relatively intact barrier function, a Franz cell diffusion assay inherently utilizes dead, enzymatically inactive skin. Thus, the results of a Franz cell assay is not necessarily clinically relevant or reflective of physiologically active skin on patients. Further work is necessary to determine whether moisturizers affects drug SC penetrance in rosacea patients.

In prior work, the investigators made method advances that overcome many of the limitations of the Franz cell assay as it relates to clinical relevance. Specifically, the investigators have established a track record of assessing drug penetrance of topically delivered medications, e.g. tazarotene, allantoin, ketoconazole, and betamethasone dipropionate, in the SC using minimally invasive D-squame tape stripes of human subjects in combination with liquid chromatography mass spectrometry (LC-MS). In these studies, the investigators are able to assess drug penetrance with physiologically relevant skin and on skin affected by the disease of interest. Therefore, the methods the investigators propose for assessing metronidazole SC penetrance in the presence of moisturizers is now established as an efficient and reliable method for quantitating drug in the SC in a minimally invasive and clinically relevant context.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, non-pregnant individual 18+ years of age;
2. Subjects willing to allow a series of tape pieces to be pressed and removed from their faces over an 4 hour period;
3. Subjects can remain calm and quiet at the research facility for 6 hours;
4. Subjects in general good health as determined from a medical history;
5. Subjects must read and sign the informed consent form after the nature of the study has been fully explained.

Exclusion Criteria:

1. Subjects with known allergies or sensitivities to ingredients contained in the test products;
2. Subjects with an allergy to latex or adhesives;
3. Subjects with excessive visible sun damage on the face, such that the dermatologist investigator considers the subject unsuitable for study entry;
4. Subjects with skin growths or other issues on the face that could interfere with the tape sampling;
5. Subjects who are currently participating in any other clinical study (i.e., dermal patch, use tests, investigational drug or devices, etc.);
6. Subjects viewed by the investigator as not being able to complete the study;
7. Subjects unwilling to refrain from using any type of lotion, medication, or other topical product to the face for a set amount of time prior to the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2024-09-03 (Actual); Primary Completion 2025-11-04 (Actual); Study Completion 2025-11-04 (Actual)

PRIMARY OUTCOMES:
Metronidazole penetrance through the stratum corneum (SC) | 1 hours and 4 hours post metronidazole application
  Metronidazole stratum corneum penetrance will be ascertained with LC-MS (liquid chromatography-mass spectrometry). Tape strips (x5) will be collected at the 1 hour and 4 hour time points post application of metronidazole.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew M Draelos, MD PhD, Principal Investigator — Duke University; John Murray, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thiboutot D, Anderson R, Cook-Bolden F, Draelos Z, Gallo RL, Granstein RD, Kang S, Macsai M, Gold LS, Tan J. Standard management options for rosacea: The 2019 update by the National Rosacea Society Expert Committee. J Am Acad Dermatol. 2020 Jun;82(6):1501-1510. doi: 10.1016/j.jaad.2020.01.077. Epub 2020 Feb 7. PMID 32035944
- [Background] Gallo RL, Granstein RD, Kang S, Mannis M, Steinhoff M, Tan J, Thiboutot D. Rosacea comorbidities and future research: The 2017 update by the National Rosacea Society Expert Committee. J Am Acad Dermatol. 2018 Jan;78(1):167-170. doi: 10.1016/j.jaad.2017.06.150. No abstract available. PMID 29102687
- [Background] Del Rosso JQ, Lehman PA, Raney SG. Impact of order of application of moisturizers on percutaneous absorption kinetics: evaluation of sequential application of moisturizer lotions and azelaic acid gel 15% using a human skin model. Cutis. 2009 Mar;83(3):119-24. PMID 19363903
- [Background] Draelos ZD, Draelos MM, Steele F, Georgiou M, Praestegaard M. Enhanced Skin Deposition of Betamethasone Dipropionate from a Novel Formulation and Drug Delivery Technology. Dermatol Ther (Heidelb). 2023 Aug;13(8):1763-1771. doi: 10.1007/s13555-023-00959-3. Epub 2023 Jun 23. PMID 37351830
- [Background] Draelos ZD, Draelos MM. Development of a Tape-Stripping Liquid Chromatography-Mass Spectrometry Method for Evaluating Skin Deposition of Topical Tazarotene. J Drugs Dermatol. 2021 Oct 1;20(10):1105-1111. doi: 10.36849/JDD.6211. PMID 34636513
- [Background] Gether L, Overgaard LK, Egeberg A, Thyssen JP. Incidence and prevalence of rosacea: a systematic review and meta-analysis. Br J Dermatol. 2018 Aug;179(2):282-289. doi: 10.1111/bjd.16481. Epub 2018 May 31. PMID 29478264
- [Background] Turpeinen M. Absorption of hydrocortisone from the skin reservoir in atopic dermatitis. Br J Dermatol. 1991 Apr;124(4):358-60. doi: 10.1111/j.1365-2133.1991.tb00597.x. PMID 2025556
- [Background] Danby SG, Draelos ZD, Gold LFS, Cha A, Vlahos B, Aikman L, Sanders P, Wu-Linhares D, Cork MJ. Vehicles for atopic dermatitis therapies: more than just a placebo. J Dermatolog Treat. 2022 Mar;33(2):685-698. doi: 10.1080/09546634.2020.1789050. Epub 2020 Jul 16. PMID 32654550
- [Background] Ghadially R, Halkier-Sorensen L, Elias PM. Effects of petrolatum on stratum corneum structure and function. J Am Acad Dermatol. 1992 Mar;26(3 Pt 2):387-96. doi: 10.1016/0190-9622(92)70060-s. PMID 1564142
- [Background] Brand RM, Charron AR, Sandler VL, Jendrzejewski JL. Moisturizing lotions can increase transdermal absorption of the herbicide 2,4-dichlorophenoxacetic acid across hairless mouse skin. Cutan Ocul Toxicol. 2007;26(1):15-23. doi: 10.1080/15569520601182791. PMID 17464745
- [Background] Huh Y, Lee DH, Choi D, Lim KM. Effect of Cosmetics Use on the In Vitro Skin Absorption of a Biocide, 1,2-Benzisothiazolin-3-one. Toxics. 2022 Feb 24;10(3):108. doi: 10.3390/toxics10030108. PMID 35324733
- [Background] Feldmann RJ, Maibach HI. Regional variation in percutaneous penetration of 14C cortisol in man. J Invest Dermatol. 1967 Feb;48(2):181-3. doi: 10.1038/jid.1967.29. No abstract available. PMID 6020682
- [Background] Tipthara P, Kobylinski KC, Godejohann M, Hanboonkunupakarn B, Roth A, Adams JH, White NJ, Jittamala P, Day NPJ, Tarning J. Identification of the metabolites of ivermectin in humans. Pharmacol Res Perspect. 2021 Feb;9(1):e00712. doi: 10.1002/prp2.712. PMID 33497030
- [Background] Vanol PG, Sanyal M, Shah PA, Shrivastav PS. Quantification of metronidazole in human plasma using a highly sensitive and rugged LC-MS/MS method for a bioequivalence study. Biomed Chromatogr. 2018 Aug;32(8):e4242. doi: 10.1002/bmc.4242. Epub 2018 Apr 22. PMID 29572903